CLINICAL TRIAL: NCT01922388
Title: Early Versus Late Application of Subthalamic Deep Brain Stimulation to Parkinson's Disease Patients With Motor Complications: a Multicentre, Prospective and Observational Study
Brief Title: Early Versus Late Application of STN DBS to PD Patients With Motor Complications
Acronym: ELASS
Status: Completed | Type: Observational
Sponsor: Chen Ling (Other)
Collaborators: Prince of Wales Hospital, Shatin, Hong Kong (Other); Shenzhen Second People's Hospital (Other)
Responsible Party: Sponsor-Investigator, Chen Ling, MD, PhD, First Affiliated Hospital, Sun Yat-Sen University
Organization: First Affiliated Hospital, Sun Yat-Sen University (Other)
Other Study IDs: [2013]19
Record Dates: First submitted 2013-08-08; First posted 2013-08-14 (Estimated); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Parkinson Disease
Keywords: Parkinson disease; deep brain stimulation; subthalamic nucleus; motor complication; quality of life
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Early Motor Complication: This group is composed of PD patients with motor complications of 3 years or less. All subjects receive bilateral deep brain stimulation of the subthalamic nucleus and best medical treatment.
  Interventions: Device: Bilateral deep brain stimulation of the subthalamic nucleus
- Late Motor Complication: This group is composed of PD patients with motor complications of more than 3 years. All subjects receive bilateral deep brain stimulation of the subthalamic nucleus and best medical treatment.
  Interventions: Device: Bilateral deep brain stimulation of the subthalamic nucleus

INTERVENTIONS:
Device: Bilateral deep brain stimulation of the subthalamic nucleus
  Other Names: Activa PC or RC neurostimulator, Medtronic

SUMMARY:
Although deep brain stimulation of the subthalamic nucleus(STN DBS) has become the surgical treatment of choice for Parkinson's disease(PD), a consensus on the timing of surgery is lacking. This study is intended to demonstrate that early, compared with delayed, introduction of STN DBS is more beneficial for PD patients who have developed motor complications.

DETAILED DESCRIPTION:
In this prospective study, 200 PD patients will be recruited for STN DBS over three years, including 133 with motor complications existing for more than three years (late complication group) and 67 less than three years (early complication group). To make a comparison of therapeutic efficacy between the two groups, motor and non-motor symptoms will be assessed using specific rating scales and questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic Parkinson's Disease with good response to levodopa(i.e. more than 30% improvement in the MDS-UPDRS Part III score after an acute levodopa challenge)
* Presence of fluctuations and/or dyskinesias
* Age ranging from 18 to 75 years old
* Normal brain MRI
* Absence of dementia (Mini Mental State Examination ≥ 26)
* Absence of severe psychiatric diseases
* Written informed consent

Exclusion Criteria:

* Presence of severe metabolic diseases
* Severe cardiac/respiratory/renal/hepatic diseases
* Secondary parkinsonism or multiple system atrophy
* Illiteracy or insufficient language skills to complete the questionnaires
* Poor compliance and unreasonable expectation
* Women who are pregnant or breast feeding
* Simultaneous participation in another clinical trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population are PD Patients with motor complications and an intention of receiving DBS.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2022-12 (Actual); Study Completion 2022-12 (Actual)

PRIMARY OUTCOMES:
Changes in 39-item Parkinson's disease questionnaire (PDQ-39) scores | From baseline to 4 years
  Quality of life

SECONDARY OUTCOMES:
Changes in Movement Disorder Society-sponsored revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part III scores | From baseline to 4 years
  Motor function
Changes in time spent in the "on" state without troubling dyskinesia based on Parkinson's disease home diary | From baseline to 4 years
  Good "on" time
Changes in MDS-UPDRS patient questionnaire (Part I B and Part II) scores | From baseline to 4 years
  Motor and non-motor experiences of daily living
Severe adverse effects | From baseline to 4 years
  Safety profile

CONTACTS AND LOCATIONS:
Overall Officials: Ling Chen, MD, PhD, Principal Investigator — First Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- the First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Jiang L, Poon WS, Moro E, Xian W, Yang C, Zhu XL, Gu J, Cai X, Liu J, Mok V, Liu Y, Xu S, Guo Q, Chen W, Chen L. Early versus Late Application of Subthalamic deep brain Stimulation to Parkinson's disease patients with motor complications (ELASS): protocol of a multicentre, prospective and observational study. BMJ Open. 2017 Nov 16;7(11):e018610. doi: 10.1136/bmjopen-2017-018610. PMID 29150478